CLINICAL TRIAL: NCT04375488
Title: Effect Of Postoperative Inspiratory Muscle Training And Strength Exercise Training On Functional Capacity, Quality of Life, Respiratory Functions, Respiratory Muscle Strength And Endurance in Bariatric Surgery Patients
Brief Title: Effect Of Strength Exercise on Respiratory Parameters, and Functional Capacity in Bariatric Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVUtacar01
Record Dates: First submitted 2020-04-17; First posted 2020-05-05 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Obesity, Morbid
Keywords: bariatric surgery; inspiratory muscle strength; respiratory muscle endurance; functional capacity; peripheral muscle strength; quality of life; resistance exercise training; 6 - Minute Walk Test
MeSH Terms: conditions — Obesity, Morbid | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Exercise Training Group (Experimental): Resistance exercise training for 8 major muscle groups and 150 min per week walking suggestions were given
  Interventions: Other: Resistance Exercise Training
- Inspiratory Muscle Training Group (Experimental): Resistance exercise training for 8 major muscle groups and inspiratory muscle strength training and 150 min per week walking suggestions were given
  Interventions: Other: Resistance Exercise Training; Other: Inspiratory Muscle Training
- Control Group (No Intervention): 150 min per week walking suggestions were given.

INTERVENTIONS:
Other: Resistance Exercise Training — 60 minutes resistance exercise training for 8 major muscle groups (quadriceps, hamstring, biceps, triceps, pectoralis major, gluteus medius , gluteus maximus, middle part of deltoid) for 8 weeks, 3 times per week
  Arms: Inspiratory Muscle Training Group; Resistance Exercise Training Group
Other: Inspiratory Muscle Training — with % 30 of MIP, 20 minutes inspiratory muscle training for 8 weeks, 3 times per week
  Arms: Inspiratory Muscle Training Group

SUMMARY:
The aim of the investigator's study is to investigate whether postoperative inspiratory muscle training and resistance exercise training has an effect on functional capacity, respiratory functions, respiratory muscle strength and endurance in patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
Obesity is an important health problem that can affect the entire organ and system of the body, leading to various disorders and even death. The fact that BMI is over 40 kg / m2 is defined as morbid obesity. The most effective treatment step in morbid obesity is bariatric surgery.

The impairment of inspiratory muscle function related to obesity is associated with increased lung elastic load, excessive lengthening in the abdominal muscles, and dissolution of the diaphragm, leading to inspiratory muscle weakness and insufficiency. The decrease in its endurance is explained by the decrease of glycogen synthase activity in skeletal muscles. It was found that there was less decrease in the inspiratory muscle training patients whose MIP values were measured before bariatric surgery compared to those who could not do MIP values after surgery.

Respiratory functions due to obesity are impaired due to restrictive mass increase in chest wall, tendency to breathe in low lung volumes and the effect of fat distribution on pleural pressure. Total lung volume, expiratory reserve volume (ERV), reserve volume (RV), vital capacity (VC), functional residual capacity (FRC), FVC, and FEV1 values are low.

After bariatric surgery, patients' muscle strength decreased. In particular, there was a decrease in muscle strength in quadriceps, hamstring, biceps, triceps. The decrease in muscle strength after surgery has been associated with a decrease in muscle mass. It was stated that patients who did not exercise after surgery lost 7.6 kg of muscle, which was 29.7% of the total lost body weight. Resistance exercises performed after bariatric surgery have a positive impact on patients' muscle strength and functional capacity.

Obesity causes a decrease in functional capacity. Increased step width, reduced walking speed and step length are shown for the main reasons. Decreased inspiratory muscle strength in patients undergoing surgery causes weakness in peripheral muscles. This weakness in peripheral muscles also reduces the functional capacity of patients. Inspiratory muscle training studies increase the functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Having a body mass index (BMI) ≥40kg / m2 or
* (BMI) ≥35kg/m2 and at least one concomitant disease associated with obesity
* To participate regularly in treatment

Exclusion Criteria:

* Using assistive device while walking
* Lung infection in the past 1 month
* Chronic obstructive pulmonary disease (COPD)
* Having an orthopedic, neurological disease that will prevent him/her from exercising
* Uncontrollable hypertension
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 3 months
  Respiratory Function Test
Forced Expiratory Volume in 1 second (FEV1) | 3 months
  Respiratory Function Test
FEV1/FVC | 3 months
  Respiratory Function Test
Peak Expiratory Flow (PEF) | 3 months
  Respiratory Function Test
Forced expiratory flow over the middle one half of the FVC (FEF25-75%) | 3 months
  Respiratory Function Test
maximum inspiratory pressure (MIP) | 3 months
  Respiratory Muscle Strength Test
Maximal Voluntary Ventilation | 3 months
  Respiratory Muscle Endurance Test
Hand-held Dynamometer | 3 months
  Dynamic Muscle Strength Test
5 times sit to stand test | 3 months
  Mobility Test
6 minutes walking test | 3 months
  functional capacity test
Quality of Life Scale Specific for Obese Persons | 3 months
  Quality of Life
maximum expiratory pressure (MEP) | 3 months
  Respiratory Muscle Strength Test
Hand grip dynamometer | 3 months
  Static Peripheral Muscle Strength Test

CONTACTS AND LOCATIONS:
Overall Officials: Alis Kostanoğlu, Study Chair — Assistant professor
Locations (1):
- Bezmialem Vakıf Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No